CLINICAL TRIAL: NCT00363740
Title: Clinical Evaluation of GW685698 for Seasonal Allergic Rhinitis -A Placebo-controlled Study to Determine the Non-inferiority of GW685698 Over Fluticasone Propionate Using a Double-blind Manner-
Brief Title: Study of GW685698X In Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR100652
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: GW685698X; allergic rhinitis; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: GW685698X Aqueous Nasal Spray

SUMMARY:
This study was designed to compare the efficacy and safety of an investigational nasal spray compared with placebo nasal spray and commonly used drug in the treatment of seasonal allergic rhinitis. Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. The focus of this study, seasonal allergic rhinitis (SAR), is one type of allergic rhinitis that is triggered by the pollen from trees, grasses, and weeds. Typical symptoms are sneezing, nasal congestion and pruritus, rhinorrhea, and pruritic, watery, red eyes.

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Outpatient
* Diagnosis of seasonal allergic rhinitis with symptoms
* Able to comply with study procedures

Exclusion Criteria:

* Significant concomitant medical condition
* Use of corticosteroids/allergy medications
* Laboratory abnormality
* Positive pregnancy test
* Allergy to any component of investigational product

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-02-19; Primary Completion 2005-04-01 (Actual); Study Completion 2005-04-13 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline over the entire treatment period in three total nasal symptom scores.

SECONDARY OUTCOMES:
Mean change from baseline over the entire treatment period in four total nasal symptom scores.
Mean change from baseline over the entire treatment period in individual total nasal symptom scores.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site